CLINICAL TRIAL: NCT04332029
Title: Smoking Cessation Treatment for Smokers With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government); State Research Agency, Spain (Other Government); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Gloria García Fernández, PhD, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCIU-19-RTI2018-101465-A-I00
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco Use Disorder, Overweight, Obesity, Eating Disorders
MeSH Terms: conditions — Tobacco Use Disorder; Overweight; Obesity; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to each of the two treatment conditions in accordance with a computer-generated randomization list. The treatment conditions will be actively running in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT + WGP + CM (Experimental): The experimental intervention includes three components: 1) Cognitive Behavioral Treatment (CBT) for gradual smoking cessation; 2) Weight Gain Prevention module (WGP) and; 3) Contingency Management (CM) procedure reinforcing tobacco abstinence.
  Interventions: Behavioral: CBT + WGP + CM
- CBT + WGP (Active Comparator): The active comparator will include only the first two components of the experimental intervention: 1) Cognitive Behavioral Treatment (CBT) for gradual smoking cessation and 2) Weight Gain Prevention module (WGP).
  Interventions: Behavioral: CBT + WGP

INTERVENTIONS:
Behavioral: CBT + WGP + CM — The intervention will be implemented in 8-week group-based sessions and includes: 1) A Cognitive Behavioral Treatment (CBT) for smoking cessation with quit date occurring at sixth session. Patients will be asked to reduce their nicotine intake gradually (i.e., 20% each week); 2) A Weight Gain Prevention module (WGP) which will consist on providing CBT and Dialectical-Behavioral Therapy (DBT) techniques targeting weight stability and associated disordered eating, and 3) a Contingency Management procedure reinforcing smoking abstinence. This component will consist on providing vouchers to reinforce abstinence contingent on biochemical verification. The schedule will incorporate an increasing magnitude of reinforcement.
  Arms: CBT + WGP + CM
Behavioral: CBT + WGP — The intervention will be implemented in 8-week group-based sessions and will include only the first two components of the experimental intervention: 1) A Cognitive Behavioral Treatment (CBT) for smoking cessation with quit date occurring at sixth session. Patients will be asked to reduce their nicotine intake gradually (i.e., 20% each week); 2) A Weight Gain Prevention module (WGP) which will consist on providing CBT and Dialectical-Behavioral Therapy (DBT) techniques targeting weight stability and associated disordered eating.
  Arms: CBT + WGP

SUMMARY:
This study aims to developed an empirically validated psychological intervention protocol for smoking cessation among individuals with excess weight. Participants will be assigned to one of the two following conditions: 1) Cognitive-Behavioral Treatment (CBT) for smoking cessation + a Weight Gain Prevention module (WGP); 2) the same treatment alongside Contingency Management (CM) for smoking abstinence.

The main goals are: 1) to assess smoking abstinence rates in each condition at post-treatment and one, three, six and twelve month follow-ups, 2) to assess the effect of treatment conditions and abstinence on weight at each assessment point, 3) to analyze the potential moderating effect of individual variables: socio-demographic characteristics, severity of nicotine dependence and demand, disordered eating, impulsivity and emotional regulation.

DETAILED DESCRIPTION:
Smoking rates are quite high among overweight or obese population. In this regard, smokers with excess weight use to report fear to quit due to post-cessation weight gain concerns, the presence of disordered eating (binge eating and emotional eating) before or during the quitting process, weight increase, relapse risk, risk of metabolic syndrome, obesity or diabetes and cardiovascular risk factors. Despite previous efforts, research is still required to assess the course of eating-related problems in smoking cessation, the impact of smoking on the onset and development of psychological and medical issues and, particularly, it is necessary to perform studies to assess the efficacy of psychological interventions for smoking cessation among individuals with excess weight. Prior evidence showed that Contingency Management (CM) techniques are adequate to reduce tobacco use and perform better than other interventions and control conditions. Nevertheless, there is a lack of research exploring the effectiveness of CM for overweight or obese smokers.The primary aim of this clinical trial is to yield data on the effectiveness of a psychological intervention for smoking cessation among individuals with excess weight. Participants will be assigned to one of the two following conditions: 1) Cognitive-Behavioral Treatment (CBT) for gradual smoking cessation + a Weight Gain Prevention module (WGP) for weight stability; 2) the same treatment alongside Contingency Management (CM) for smoking abstinence. In view to assure adequate power for achieving statistical significance, investigators carried out a priori power analysis by using the G*Power 3.1. An estimated sample size of 120 participants would detect a medium effect size (Cohen's d = 0.3, with power (1-β) set at 0.97 and α = 05).The primary analyses derived from this clinical trial will be conducted using Statistical Package for the Social Science (SPSS) version 24 for Windows. A set of descriptive and frequency analyses will be carried out with regard to participants' characteristics. Comparisons between treatment groups in both baseline characteristics and treatment outcomes will be conducted using a set of chi-square tests for categorical variables and t-tests (two-tailed) for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 or over.
* Having smoked 10 or more cigarettes/day within the last year.
* Meeting the diagnostic criteria for nicotine dependence according to the Diagnostic and Statistical Manual of Mental Disorders-5th ed. (American Psychiatric Association 2013).
* Having overweight or obesity (BMI above 25)

Exclusion Criteria:

* Not being able to attend the entire treatment.
* Being currently receiving other psychological/pharmacological treatment for smoking cessation or weight control
* Being diagnosed with a current severe psychiatric disorder, eating disorder other than Binge-Eating Disorder or Substance Use Disorder other than nicotine.
* Being pregnant, lactating or in the postpartum period
* Have any health condition that requires a specialized diet or aﬀected eating
* Participants must not be taking a medication that impacts weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in Smoking abstinence | Through Study Completion: End-of-treatment (8-week), 1, 3, 6 and 12 month follow-up
  Abstinence is defined as achieving a period of at least 24 hours of abstinence (end-of-treatment) or not smoking since the prior last 7 days. Abstinence is assessed by means of carbon monoxide (CO) and cotinine samples.
Changes in Continuous smoking abstinence | Through Study Completion: End-of-treatment (8-week), 1, 3, 6 and 12 month follow-up.
  Abstinence is defined as no smoking (not even a puff) since the participant´s quit day. Abstinence is assessed by means of carbon monoxide (CO) and cotinine samples
Weight Change | Through Study Completion: End-of-treatment (8-week), 1, 3, 6 and 12 month follow-up
  At all measurement visits, weight will be recorded in kilograms. Weight will be measured on a calibrated digital scale in duplicate, with the participant wearing light clothing and no shoes.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Unit of Addictive Behaviors. Faculty of Psychology. University of Oviedo., Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia-Fernandez G, Krotter A, Garcia-Perez A, Aonso-Diego G, Secades-Villa R. Pilot randomized trial of cognitive-behavioral treatment plus contingency management for quitting smoking and weight gain prevention among smokers with overweight or obesity. Drug Alcohol Depend. 2022 Jul 1;236:109477. doi: 10.1016/j.drugalcdep.2022.109477. Epub 2022 Apr 29. PMID 35525238